CLINICAL TRIAL: NCT06150495
Title: Glycemic Control and Retinal Microvascular Changes in Type 2 Diabetes Mellitus Patients Without Clinical Retinopathy
Brief Title: Glycemic Control and Retinal Microvascular Changes
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: IRB no. 2021-06-029
Record Dates: First submitted 2023-11-12; First posted 2023-11-29 (Actual); Last update posted 2023-11-29 (Actual); Status verified 2023-11

CONDITIONS: Diabetic Retinopathy; Neurodegeneration; Blood Sugar; High
MeSH Terms: conditions — Diabetic Retinopathy; Nerve Degeneration; Hyperglycemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Healthy control: The controls included patients without DM who presented for regular ophthalmic examination.
- intensive control (IC) group: The mean HbA1c level was calculated during the 12 months prior to the OCT and OCTA. Based on the mean HbA1c level, T2DM patients were divided into intensive control (IC; mean HbA1c ≤ 7.0%) and moderate control (MC; mean HbA1c > 7.0%) groups
- moderate control (MC) group: The mean HbA1c level was calculated during the 12 months prior to the OCT and OCTA. Based on the mean HbA1c level, T2DM patients were divided into intensive control (IC; mean HbA1c ≤ 7.0%) and moderate control (MC; mean HbA1c > 7.0%) groups

SUMMARY:
The goal of this prospective, observational study is to compare in the association of glycemic control and retinal microvascular changes in patients with type 2 diabetes mellitus (T2DM) without diabetic retinopathy (DR).

The main question it aims to answer are:

• Do degenerative changes in retinal microvasculature or nerves depend on glycemic control even before diabetic retinopathy is detected?

Participants will receive an annual routine comprehensive examination including ultra-widefield fundus photography, spectral domain optical coherence tomography (OCT), and swept-source optical coherence tomography angiography (OCTA).

ELIGIBILITY:
Inclusion Criteria:

* The study included 30-70-year-old patients with T2DM without known DR at baseline who underwent regular screening for DR at the department of ophthalmology.
* Who underwent regular checkups for DR between January 2019 and August 2022 at Dongguk University Ilsan Hospital.
* The controls included patients without DM who presented for regular ophthalmic examination.

Exclusion Criteria:

* patients with a history of retinal or choroidal diseases (i.e., age-related macular degeneration, retinal vein occlusion, uveitis, retinal detachment, and central serous chorioretinopathy), glaucoma, or optic neuropathy
* patients with neurodegenerative diseases, such as Parkinson's disease and dementia.

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study included 30-70-year-old patients with T2DM without known DR at baseline who underwent regular screening for DR at the department of ophthalmology. The controls included patients without DM who presented for regular ophthalmic examination. One eye each of DM patients and controls was included in the study. The eye without significant ocular disease was selected from both eyes; if both eyes were eligible, the right eye was selected. The participants underwent comprehensive ophthalmic examination, including best-corrected visual acuity assessment using the Snellen chart, slit-lamp biomicroscopy, dilated fundus examination, ultra-widefield fundus photography, spectrum-domain OCT, and SS-OCTA. Patients with T2DM were included in the study after a retinal specialist confirmed absence of signs of DR on clinical examination and ultra-wide fundus photography.
Sampling Method: Non-Probability Sample
Enrollment: 259 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2022-08-31 (Actual); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
The foveal avascular zone (FAZ) area (mm^2) | Upon initial registration and through study completion, an average of 1 year
  FAZ was defined as the avascular area in the foveal center.
central foveal retinal thickness (um) and macular ganglion cell-inner plexiform layer (GC-IPL) thickness (um) | Upon initial registration and through study completion, an average of 1 year
  Retinal layer thickness were calculated automatically using the bundled software
Retinal vessel density (VD, %) | Upon initial registration and through study completion, an average of 1 year
  The VD (%) was calculated using the following formula: VD (%) = vascular area (pixel) / (total area - FAZ area) (pixel) × 100.

CONTACTS AND LOCATIONS:
Locations (1):
- Dongguk University Ilsan Hospital, Goyang-si, Republic of Korea, South Korea

IPD SHARING:
Plan to Share IPD: Undecided